CLINICAL TRIAL: NCT01596972
Title: The Role of a Semi-Quantitative Urine Pregnancy Test and Pregnancy Questionnaire After Uterine Evacuation for Undesired Pregnancy of Uncertain Location: A Pilot Randomized Controlled Trial
Brief Title: The Role of a Semi-Quantitative Urine Pregnancy Test and Pregnancy Questionnaire After Uterine Evacuation for Undesired Pregnancy of Uncertain Location
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2012P000576
Record Dates: First submitted 2012-05-08; First posted 2012-05-11 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Follow-up After Uterine Evacuation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Serum quantitative urine pregnancy test (Experimental): uterine evacuation follow-up consisting of an at-home, self-administered SQ-UPT and standardized pregnancy symptom questionnaire in 1 week
  Interventions: Device: dBest semi-quantitative urine pregnancy test
- serum hCG (No Intervention): follow-up consisting of a 1 week return visit and serum hCG plus standardized pregnancy symptom questionnaire

INTERVENTIONS:
Device: dBest semi-quantitative urine pregnancy test — The dBest® semi-quantitative urine pregnancy test (Figure 2) is a graduated urine pregnancy test with five different levels of sensitivity: 25 IU/L, 100 IU/L, 500 IU/L, 2000 IU/L, 10000 IU/L. The test detects the level of serum hCG that corresponds to the range between that level and the level above it, i.e. the test would be positive at 500 if the hCG was either 501 or 1999. The tool was validated in a US sample of 196 women, where there was a correlation of 69% between urine hCG and serum hCG. Furthermore, the test had a 10% false negative rate (i.e. recording a level two gradations below the serum level) and a 6% false positive rate (i.e. recording a level two gradations above the serum level)
  Arms: Serum quantitative urine pregnancy test

SUMMARY:
The primary aim of this study is to determine if a self-administered semi-quantitative urine pregnancy test and telephone pregnancy symptom questionnaire can reduce the percentage of women with a complete uterine evacuation who require a clinic or lab visit to confirm completion.

The investigators hypothesize that women with complete uterine evacuation will be less likely to require a follow-up clinic or lab visit by using a standardized pregnancy questionnaire and home SQ-UPT, than by using serum hCG as the objective measure of completion.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older with an undesired pregnancy < 6 weeks gestation
* Women with a positive urine pregnancy test
* Proficiency in English
* Working phone and subject willing to be contacted by phone.
* Agreeing to surveys regarding demographics, follow-up preferences, and satisfaction with assigned follow-up method

Exclusion Criteria:

* Women with presence of a yolk sac or crown rump length visualized on ultrasound
* Women with a gestational sac greater than 13mm [11]
* High Suspicion for ectopic pregnancy

  o Sign: Concerning adnexal mass seen on ultrasound in conjunction with pelvic pain and/or vaginal spotting
* Hemodynamic instability

  o Signs: heavy vaginal bleeding, hypotension, tachycardia
* Pelvic Infection

  o Signs: pain or fever
* Medical conditions that contraindicate uterine evacuation according to PPLM clinic policy

  o These include but are not limited to: a bleeding disorder or anticoagulation, significant cardiac disease, renal or liver failure, IUD in situ that cannot be removed
* Unwilling or unable to comply with study follow-up procedures
* Being in a situation where receiving phone calls or additional contact with research staff may endanger the privacy or safety of the subject (e.g. situations of domestic violence or abuse)
* Inability to give informed consent
* Previous participation in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, MPH, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 2012-March 2013 Outpatient clinic
Period: Overall Study
Arm/Group | Serum Quantitative Urine Pregnancy Test | Serum hCG
Started | 25 | 26
Completed | 24 | 12
Not Completed | 1 | 14
Not completed — Physician Decision | 1 | 9
Not completed — Lost to Follow-up | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Serum Quantitative Urine Pregnancy Test | Serum hCG | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (5) | 25 (5) | 25 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — The numbers below report self-described RACE of participants. Additionally, though, 3 participants in the Serum HCG arm and 5 participants in the serum quantitative urine pregnancy test arm also self-identified as having a Hispanic Ethnicity.
  participants
    White/European American | 14 | 14 | 28
    Black/African American | 5 | 3 | 8
    Asian | 2 | 4 | 6
    Multiracial | 2 | 4 | 6
    Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Women in Each Group Who Require a Return Visit to the Clinic for a Serum hCG Measurement, Ultrasound or Clinical Examination at One Week to Confirm Complete Evacuation
Time Frame: 1 week
Population: The number of participants analyzed in the serum hCG arm were the number of participants who started in this arm minus the number who were discontinued from the study per MD decision (total N in analysis was therefore 17).
Measure: Number; unit: participants
Arm/Group | Serum Quantitative Urine Pregnancy Test | Serum hCG
Number analyzed (Participants) | 24 | 17
participants | 3 | 17

2. Secondary Outcome: Patient Compliance With Each Follow-up Method
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Serum Quantitative Urine Pregnancy Test | Serum hCG
Number analyzed (Participants) | 24 | 17
participants | 24 | 12

3. Secondary Outcome: Patient Satisfaction With Each Follow-up Method
Description: Patient satisfaction with each follow-up method was assessed with the following survey questions:
  How satisfied are you with [name of follow-up method]? (very satisfied, satisfied, neutral, unsatisfied, very unsatisfied)
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | Serum Quantitative Urine Pregnancy Test | Serum hCG
Number analyzed (Participants) | 24 | 17
participants | 22 | 6

ADVERSE EVENTS:
Arm/Group | Serum Quantitative Urine Pregnancy Test | Serum hCG
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No